CLINICAL TRIAL: NCT00800319
Title: ALK33-001: A Phase 1 Study of the Pharmacokinetics of RDC-0313 Administered to Healthy Adults
Brief Title: ALK33-001: A Study of RDC-0313 Administered to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK33-001
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; Opioid antagonist; RDC-0313
MeSH Terms: conditions — Alcoholism | interventions — ALKS-33

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- RDC-0313, 5mg (Experimental): 5 mg of RDC-0313; single dose
  Interventions: Drug: RDC-0313
- RDC-0313, 15 mg (Experimental): 15 mg RDC-0313; single dose
  Interventions: Drug: RDC-0313
- RDC-0313, 25mg (Experimental): 25 mg RDC-0313; single dose
  Interventions: Drug: RDC-0313
- RDC-0313, 50 mg (Experimental): 50 mg RDC-0313; single dose
  Interventions: Drug: RDC-0313
- RDC-0313, 75 mg (Experimental): 75 mg RDC-0313; single dose
  Interventions: Drug: RDC-0313
- Placebo (Placebo Comparator): volume-match placebo; single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RDC-0313 — Oral solution given in 5, 15, 25, 50, and 75 mg single doses
  Arms: RDC-0313, 15 mg; RDC-0313, 25mg; RDC-0313, 50 mg; RDC-0313, 5mg; RDC-0313, 75 mg
Drug: Placebo — Volume matched placebo; oral solution; single dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the pharmacokinetics, safety, and tolerability of RDC-0313 following oral administration.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, ascending dose, placebo controlled study. Dosing sequences will consist of 5 administrations of an oral solution of either ascending doses of RDC-0313 or volume-match placebo. Dosing of cohorts will be staggered to allow a blinded safety review to occur prior to dosing the next cohort. Subjects will be admitted to the facility the morning before each dose, and will be required to fast overnight prior to study drug administration. They will be discharged from the facility after the 36-hour postdose assessments are completed.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years of age
* Body mass index of 19-30 kg/m2 at screening
* If subject is female and of childbearing potential, she must agree to use an acceptable method of contraception
* If subject is male, he must agree to reduce the risk of a female partner becoming pregnant

Exclusion Criteria:

* Pregnancy and/or currently breastfeeding
* Clinically significant medical condition or observed abnormalities
* Clinically significant illness within 30 days of the first study drug administration
* History of opioid dependence
* Positive urine toxicological screen for marijuana, cocaine, amphetamines, opioids, barbiturates, and benzodiazepines
* Positive resolut for any serology test performed at screening
* Use of alcohol-, caffeine-, or xanthine-containing products
* Tobacco use within 90 days before the first study drug administration
* Participation in a clinical trial within 30 days before screening
* Requirement of a special diet other than vegetarian, or significant food allergy or intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentrations (Cmax) of RDC-0313 | 12 weeks

SECONDARY OUTCOMES:
Clinically significant abnormal laboratory findings | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip T. Leese, MD, Principal Investigator — Quintiles Phase One Services
Locations (1):
- Quintiles Phase One Services, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Turncliff R, DiPetrillo L, Silverman B, Ehrich E. Single- and multiple-dose pharmacokinetics of samidorphan, a novel opioid antagonist, in healthy volunteers. Clin Ther. 2015 Feb 1;37(2):338-48. doi: 10.1016/j.clinthera.2014.10.001. Epub 2014 Oct 29. PMID 25456560